CLINICAL TRIAL: NCT02375815
Title: The Statin Choice Implementation Project: Phase 1
Brief Title: Statin Choice Decision Aid Implementation First Phase
Acronym: SCIP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Victor Montori, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-006048
Record Dates: First submitted 2015-02-16; First posted 2015-03-03 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Factor Risk
Keywords: statin; decision aid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Statin Choice Implementation (Experimental)
  Interventions: Other: Statin Choice Implementation

INTERVENTIONS:
Other: Statin Choice Implementation

SUMMARY:
This study is designed to answer a key question in the field of implementation science. Specifically, it seeks to determine if a proposed model for the implementation and scale-up of healthcare innovations (the AIDED model) is effective and useful. To fully evaluate the potential of this model, the investigators will conduct a multi-year study comprising 3 phases. This proposal represents the first of these phases.

ELIGIBILITY:
Subjects of the Mayo Clinic Care Network

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Effective Implementation of Statin Choice Decision Aid (SCDA), as indicated by the cumulative reach (% usage in appropriate primary care consultations) across all 3 health systems (as measured by EMR-based calculations). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor Montori, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Kootenai Health, Coeur d'Alene, Idaho
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mosaic Life Care, Saint Joseph, Missouri
  - Altru Health System, Grand Forks, North Dakota

REFERENCES:
- [Derived] Leppin AL, Boehmer KR, Branda ME, Shah ND, Hargraves I, Dick S, Elwyn G, Ting HH, Ye S, Gilles R, Abbas M, Alexander A, Montori VM. Developing a toolkit to implement the Statin Choice Conversation Aid at scale: application of a work reduction model. BMC Health Serv Res. 2019 Apr 24;19(1):249. doi: 10.1186/s12913-019-4055-8. PMID 31018840